CLINICAL TRIAL: NCT05166863
Title: Physical Performance Testing and Frailty in Prediction of Early Postoperative Course After Cardiac Surgery
Acronym: Cardiostep
Status: Active, not recruiting | Type: Observational
Sponsor: Jan Gofus, MD, PhD (Other)
Collaborators: Charles University, Czech Republic (Other)
Responsible Party: Sponsor-Investigator, Jan Gofus, MD, PhD, Deputy Chief for Science and Research, University Hospital Hradec Kralove
Organization: University Hospital Hradec Kralove (Other)
Other Study IDs: 202010 P07
Record Dates: First submitted 2021-12-08; First posted 2021-12-22 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Cardiac Surgery; Rehabilitation; Frailty; Physical Performance
Keywords: surgery, rehabilitation, frailty, performance, activity
MeSH Terms: conditions — Frailty; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Standard risk prediction models in cardiac surgery (such as EuroSCORE II or STS score) are designed to analyze solely the risk of short-term postoperative mortality. The postoperative morbidity, the ability to rehabilitate or the mid-term survival are not addressed by these means. Recently there have been some reports that addition of physical performance testing to the standard prediction models may provide prognostic value. There is a wide scale of various physical performance and frailty tests that could be used for this purpose, but they have not been confronted with each other yet. Moreover, the postoperative physical rehabilitation has not been objectively assessed in larger scale despite the significant improvement in technology.

The hypothesisis of the study is that the preoperative outcomes of physical performance and frailty testing are able to predict the patient's reconvalescence after cardiac surgery in the short- and mid-term postoperatively. The aim is to analyze a set of tests with regard to their ability to predict postoperative reconvalescence, including the objective activity assessment (using Actigraph wGT3X-BT activity tracking device). Secondarily, the investigators aim to follow the patients up to 1 year postoperatively in terms of evaluating their mid-term outcomes.

DETAILED DESCRIPTION:
Detailed description of testing performed in the exact order as in the patient:

1. Body weight and body composition (weigth of fat, weigth of muscle) measurement using bioimpendance scale Tanita BC 545N.
2. Katz Index of Independence in Activites of Daily Living performed and assessed exactly as described elsewhere.
3. Hand-grip strength test using the Kern MAP 80K1 device. Modified Southhampton protocol will be used for the measurement: Patient is sitting on a chair without side arms, the elbows are in a right angle. The patient is instructed to squeeze the device as much as possible and hold for 3 seconds. He squeezes the device with the right hand, then with the left hand. This is performed two times with each hand in total. The highest measured value is recorded.
4. 5-meter gait test. Patient is instructed to walk the 5-meter line as fast as possible and the time is being measured. This is repeated three times. Average time of the three attempts is recorded.
5. 6-minute walk test. Patient is instructed to walk without interruption for 6 minutes in the corridor of department's standard ward (exactly 36 meters long). He walks there and back repeatedly and the walked distance is calculated with regard to the number of corridors walked.
6. During the last two tests patient is wearing a pulse oxymeter (Berry BM1000C) that is connected with investigator's smartphone (either Android or iOS) through bluetooth. Eventual latent respiratory failure is recorded, defined as a drop in peripheral saturation of 4 % and more, or under 88 %.
7. Pre-defined set of laboratory blood tests: haemoglobin, creatinin, albumin, TSH, free T3, free T4.

ELIGIBILITY:
Inclusion Criteria:

* informed patient consent
* patient scheduled for an elective cardiac surgery. The following procedures are accepted: coronary artery bypass grafting (CABG) , single valve replacement (SVR), CABG + SVR, CABG + MAZE procedure, SVR + MAZE procedure
* since June 2021, patients undergoing double-valve surgery have been allowed to be included in the study to promote patients inclusion

Exclusion Criteria:

* complex cardiac surgery (except the options listed above)
* ejection fraction of the left ventricle < 30 % according to the last preoperative echocardiography
* EuroSCORE II value > 5 %
* urgent or emergent surgery
* patient unable to walk and/or perform the test
* severe dementia (due to unability to cooperate during the testing and follow-up)
* re-do surgery
* minimally invasive surgery (i.e. other than full median sternotomy)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for non-complex elective cardiac surgery at a single tertiary care cardiovascular center in the Czech Republic.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Standard postoperative measures of patient reconvalescence | Usually up to 30 days postoperatively
  To analyze the ability of preoperative physical performance and frailty tests to predict the standard postoperative measures of patient reconvalescence: length of artificial ventilation, length of stay in the intensive care unit, total postoperative hospital stay.
Objective postoperative patient activity tracking | First 4 postoperative days in the standard ward
  To analyze the ability of preoperative physical performance and frailty tests to predict the outcomes of objective postoperative patient activity tracking by the means of total number of steps taken during the first 4 days in the standard ward and total intensity of physical activity in this time period, both measured by the dedicated wearable Actigraph activity monitor.

SECONDARY OUTCOMES:
The dynamics of physical performance in the mid-term postoperatively | 1 year postoperatively
  To repeat the set of preoperative physical and frailty tests in pre-specified time intervals after the surgery: on 7th postoperative day, 3 months after the surgery and 1 year after the surgery. Thereafter, the investigators aim to evaluate the dynamics of the outcomes and eventual predictive value of the preoperative outcomes.
Mid-term postoperative mortality, major adverse events, cardiac rehospitalizations | 1 year postoperatively
  To analyze the ability of preoperative physical performance and frailty tests to predict the 1-year (mid-term) postoperative mortality, major adverse cardiac and cerebrovascular events and the risk of rehospitalizations for cardiac reasons.

CONTACTS AND LOCATIONS:
Overall Officials: Ján Gofus, MD, PhD, Principal Investigator — University Hospital Hradec Králové; Jan Vojáček, Professor, MD, PhD, Study Chair — University Hospital Hradec Králové
Locations (1):
- University Hospital Hradec Králové, Hradec Králové, Královehradecký Kraj, Czechia

IPD SHARING:
Plan to Share IPD: Undecided
The anonymized individual patient data will be shared upon a reasonable request to the principal study investigator.

REFERENCES:
- [Background] de Arenaza DP, Pepper J, Lees B, Rubinstein F, Nugara F, Roughton M, Jasinski M, Bazzino O, Flather M; ASSERT (Aortic Stentless versus Stented valve assessed by Echocardiography Randomised Trial) Investigators. Preoperative 6-minute walk test adds prognostic information to Euroscore in patients undergoing aortic valve replacement. Heart. 2010 Jan;96(2):113-7. doi: 10.1136/hrt.2008.161174. Epub 2009 Jun 28. PMID 19561363
- [Background] Afilalo J, Eisenberg MJ, Morin JF, Bergman H, Monette J, Noiseux N, Perrault LP, Alexander KP, Langlois Y, Dendukuri N, Chamoun P, Kasparian G, Robichaud S, Gharacholou SM, Boivin JF. Gait speed as an incremental predictor of mortality and major morbidity in elderly patients undergoing cardiac surgery. J Am Coll Cardiol. 2010 Nov 9;56(20):1668-76. doi: 10.1016/j.jacc.2010.06.039. PMID 21050978
- [Background] Gofus J, Vobornik M, Koblizek V, Pojar M, Vojacek J. The outcome of a preoperative one-minute sit-to-stand test is associated with ventilation time after cardiac surgery. Scand Cardiovasc J. 2021 Jun;55(3):187-193. doi: 10.1080/14017431.2020.1866771. Epub 2020 Dec 26. PMID 33356620
- [Background] Afilalo J, Lauck S, Kim DH, Lefevre T, Piazza N, Lachapelle K, Martucci G, Lamy A, Labinaz M, Peterson MD, Arora RC, Noiseux N, Rassi A, Palacios IF, Genereux P, Lindman BR, Asgar AW, Kim CA, Trnkus A, Morais JA, Langlois Y, Rudski LG, Morin JF, Popma JJ, Webb JG, Perrault LP. Frailty in Older Adults Undergoing Aortic Valve Replacement: The FRAILTY-AVR Study. J Am Coll Cardiol. 2017 Aug 8;70(6):689-700. doi: 10.1016/j.jacc.2017.06.024. Epub 2017 Jul 7. PMID 28693934
- [Background] Abdullahi YS, Salmasi MY, Moscarelli M, Parlanti A, Marotta M, Varone E, Solinas M, Sheriff RM, Casula RP, Athanasiou T. The Use of Frailty Scoring to Predict Early Physical Activity Levels After Cardiac Surgery. Ann Thorac Surg. 2021 Jan;111(1):36-43. doi: 10.1016/j.athoracsur.2020.06.029. Epub 2020 Aug 18. PMID 32818541
- [Background] Cook DJ, Thompson JE, Prinsen SK, Dearani JA, Deschamps C. Functional recovery in the elderly after major surgery: assessment of mobility recovery using wireless technology. Ann Thorac Surg. 2013 Sep;96(3):1057-61. doi: 10.1016/j.athoracsur.2013.05.092. PMID 23992697
- [Background] Joshi A, Mancini R, Probst S, Abikhzer G, Langlois Y, Morin JF, Rudski LG, Afilalo J. Sarcopenia in cardiac surgery: Dual X-ray absorptiometry study from the McGill frailty registry. Am Heart J. 2021 Sep;239:52-58. doi: 10.1016/j.ahj.2021.04.008. Epub 2021 May 4. PMID 33957101
- [Background] Hosler QP, Maltagliati AJ, Shi SM, Afilalo J, Popma JJ, Khabbaz KR, Laham RJ, Guibone K, Kim DH. A Practical Two-Stage Frailty Assessment for Older Adults Undergoing Aortic Valve Replacement. J Am Geriatr Soc. 2019 Oct;67(10):2031-2037. doi: 10.1111/jgs.16036. Epub 2019 Jun 18. PMID 31211413
- See also: Website and detailed information on the ActiGraph Activity Tracking Device — https://www.actigraph.nl/en/